CLINICAL TRIAL: NCT02002728
Title: Comparison of Early Caries Detection in Children Utilizing an Electrical Conductance Device and the Gold Standard of Visual-tactile Technique.
Status: Completed | Type: Observational
Sponsor: Ortek Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ECD0613
Record Dates: First submitted 2013-12-01; First posted 2013-12-06 (Estimated); Last update posted 2013-12-09 (Estimated); Status verified 2013-12

CONDITIONS: Dental Caries in Children

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 14 Months
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to evaluate a methodology for detecting early forming cavities in children that is more accurate and reliable than the gold standard used by dentists around the world. The new method uses an electrical current device to detect early enamel mineral loss before it can develop into a cavity. The manual gold standard is for a dentist to probe the surfaces of the teeth with a fine pick, searching for areas of defect.

ELIGIBILITY:
Inclusion Criteria:

Children whose parents authorize participation by signing a consent form. Children who attend public school only. Children in good health. Children between 6 and 9 years of age. Children with all first permanent molars erupted. All permanent first molars must not have any signs of cavitation but only one molar can have some mineral loss(e.g. white spots).

Children must show some caries in the primary molars as a sign of caries susceptibility.

-

Exclusion Criteria:

Children of parents or a guardian who do not agree to participate in the study. Children registered in private schools. Children not in good health. Children undergoing antimicrobial or antibiotic treatment. Children outside the range of age selected for the study. Children with one or more first permanent molars unerupted. Children with any cavitation in the occlusal surface of any first permanent molar.

Children who do not have a sign of dental caries in the primary molars as a sign of caries susceptibility.

Children who do not allow themselves to be examined.

-

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children ages 6 - 9 years.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2006-11; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
To compare the detection of occlusal caries lesions in the first permanent molars of Venezuelan children by electrical conductance and visual-tactile means. | 14 months from baseline assessment

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Central de Venezuela, Caracas, Venezuela, Venezuela